CLINICAL TRIAL: NCT03661697
Title: Effect of Combination Laser Treatment and Skin Brightening Topical on the Appearance of Skin Tone and Photoaging: A Pilot Study
Brief Title: Combination Versus Laser Treatment Only
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: Allergan Sales, LLC (Industry)
Responsible Party: Principal Investigator, Lisa Grunebaum, Associate Professor of Facial Plastic and Reconstructive Surgery and Dermatology, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20171006
Record Dates: First submitted 2018-09-05; First posted 2018-09-07 (Actual); Results first posted 2020-04-24 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Photoaging
Keywords: skin; sun damage; photoaging of face; skin care; laser therapy
MeSH Terms: interventions — Laser Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Lytera Arm (Experimental): 4 week washout period with skin care regimen including Lytera 2.0 followed by 2 laser treatments.
  Interventions: Device: Laser Therapy; Other: Basic Skin Care Regimen; Other: Lytera
- Laser only arm (Active Comparator): 4 week washout period with a basic skin care regimen, no Lytera 2.0, followed by 2 laser treatments.
  Interventions: Device: Laser Therapy; Other: Basic Skin Care Regimen

INTERVENTIONS:
Device: Laser Therapy — Clear and Brilliant Permea is a 1927nm fractional laser with 3 settings; low, medium, high.
  All interventions were done at low with four passes to each participant's full face.
  Other Names: Clear and Brilliant Permea (1927nm fractional)
Other: Basic Skin Care Regimen — Skin Medica brand cleanser, sunscreen, moisturizer as directed for 12 weeks
Other: Lytera — cosmeceutical serum applied to face daily for 12 weeks
  Arms: Lytera Arm

SUMMARY:
Our objective is to determine the effects of (1) basic skin care regimen + "active" (Lytera 2.0) vs. (2) basic skin care regimen only, both groups combined with laser, on the appearance of skin tone and photo-aging on the face.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult male and female patients 18 years and older
* Fitzpatrick skin types I-IV
* Has at least mild mottled skin tone of the face (score of 2 or more on a 5 point skin tone scale)
* Has at least 2 areas of the face with significant roughness, dyspigmentation, or fine lines or has all these characteristics in 1 or more areas
* Willing to refrain from using any other topical products on the face, systemic retinoids, or steroids, facial peels or other facial laser procedures throughout the duration of the study
* Willing to refrain from any cosmetic procedure including but not limited to facial surgery, dermal fillers, and neuromodulators for the duration of the study
* Willing to use only the facial skin care product regimen provided for the study
* Willing to avoid extended periods of sun exposure and the use of tanning beds during the study
* Willing to have photographs taken of the face to be used de-identified in evaluations, publications, and presentations
* For females: proof that they are not pregnant (urine pregnancy test)
* English-speaker

Exclusion Criteria:

* Has any uncontrolled systemic disease (such as autoimmune disorders and connective tissue disorders such as lupus erythematosus or Sjogren's syndrome
* Has any active infection in face
* Has history of any skin conditions that could interfere with treatment
* Has used self-tanner recently
* Is currently participating in another drug research study
* Is NOT willing to refrain from using any other topical products such as skin lightening, retinoids, alpha/beta-hydroxyl acids, salicylic acid, vitamins C or D, steroids, or antibiotics on the face or systemic retinoids, steroids, facial peels, neuromodulators, dermal fillers, facial surgery, or other facial laser procedures throughout the duration of the study
* For females: is pregnant
* Non English-speaker

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2018-10-10 (Actual); Primary Completion 2019-03-07 (Actual); Study Completion 2019-03-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Grunebaum, MD, Principal Investigator — Univeristy of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Lytera Arm: 4 week washout period with skin care regimen (facial cleanser, Lytera 2.0, TNS Ceramide Treatment Cream and Essential defense mineral shield broad spectrum SPF 35) followed by 2 laser treatments.
  Skin Care Regimen plus Lytera 2.0 and Laser Therapy: Combined
  Lytera plus Laser: two arms of study- each with different topical cosmeceutical
- Placebo Arm: 4 week washout period with a basic skin care regimen (facial cleanser, TNS Ceramide Treatment Cream and essential defense mineral shield broad spectrum SPF 35) followed by 2 laser treatments.
  Basic Skin Care Regimen Only and Laser Therapy: Not Combined
  Lytera plus Laser: two arms of study- each with different topical cosmeceutical
Period: Overall Study
Arm/Group | Lytera Arm | Placebo Arm
Started | 7 | 7
Completed | 7 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lytera Arm | Placebo Arm | Total
Number analyzed (Participants) | 7 | 7 | 14
Age, Continuous [Mean (Full Range); unit: years] | 47.43 [38 to 80] | 51.57 [23 to 68] | 49.5 [23 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 14
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 4 | 5
  Not Hispanic or Latino | 4 | 3 | 7
  Unknown or Not Reported | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 5 | 7 | 12
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change in Aesthetics
Description: Blinded evaluation using Global Aesthetic Improvement Scale (GAIS) (0=worse, 4=very much improved)
Time Frame: baseline to 12 weeks
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Lytera Arm | Placebo Arm
Number analyzed (Participants) | 7 | 7
score on a scale | 2 [1.5 to 2] | 1 [1 to 2]

2. Primary Outcome: Change in Skin Tone
Description: Change in skin tone is assessed using the Modified Pigmentation Area and Severity Index (MoPASI). MoPASI assesses three facial region variables: 1) A = % area of involvement (0 = no involvement, 6 = 90% involvement), 2) D = darkness of pigment (0=absent, 4=maximum), 3) P = pattern of involvement (0=absent, 4=maximum). Four facial regions will be assessed: Forehead (0.2A), Left Cheek and periorbital (0.3A), Right Cheek and periorbital (0.3A), Nose/Lip/Chin (0.2A). The Total score ranges from 0-48 and is calculated using the formula: MoPASI = 0.2A(D + P) + 0.3A (D+P) + 0.3A (D+P) + 0.2A (D+P). A higher score indicates higher pigmentation.
Time Frame: baseline to 12 weeks
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Lytera Arm | Placebo Arm
Number analyzed (Participants) | 7 | 7
score on a scale | -8.7 [-10.80 to -6.55] | -3.90 [-4.30 to -2.95]

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: treatment emergent
Arm/Group | Lytera Arm | Placebo Arm
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/7
Other Adverse Events (participants affected / at risk) | 2/7 | 2/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lytera Arm (N=7) | Placebo Arm (N=7)
acne (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
dryness (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-25): https://cdn.clinicaltrials.gov/large-docs/97/NCT03661697/Prot_SAP_001.pdf